CLINICAL TRIAL: NCT03815045
Title: Ultrasound Guided Diagnostic Lumbar Puncture in Neurology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An interim analysis was conducted, and no difference was found between traditional lumbar punctures and ultrasound-guided lumbar punctures. The study was subsequently terminated.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D17180
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Landmark-based lumbar puncture (Active Comparator): Landmark-based LP
  Interventions: Procedure: Landmark-based lumbar puncture
- Ultrasound-guided lumbar puncture (Active Comparator): Ultrasound-guided LP
  Interventions: Procedure: Ultrasound-guided lumbar puncture

INTERVENTIONS:
Procedure: Landmark-based lumbar puncture — Traditional landmark based lumbar puncture involves palpating spinous processes on the back and finding the inter-spinous space which is the site of needle entry to gain access to the thecal sac. Finding this space may be difficult by palpation, especially when subjects undergoing the procedure are obese, elderly, have had prior back surgery, or if the patient is positioned incorrectly.
  Arms: Landmark-based lumbar puncture
Procedure: Ultrasound-guided lumbar puncture — Ultrasound guided lumbar puncture is a novel technique being increasingly utilized by emergency physicians, pediatricians and anesthesiologists. In this technique, an ultrasound probe is used to visualize the inter-spinous space. This space can be marked on the skin as the potential point of entry. This could potentially make it easier when patient factors make it difficult to palpate and find the site of entry.
  Arms: Ultrasound-guided lumbar puncture

SUMMARY:
Subjects who are having a lumbar puncture as part of their clinical care will be randomized to either a traditional landmark based lumbar puncture or ultrasound guided lumbar puncture. The primary objective of study is to compare the success rate of obtaining CSF using Ultrasound guided technique against the Traditional Landmark based approach. Secondary objectives are to evaluate factors influencing the success or failure, patient tolerance, and a safety assessment.

DETAILED DESCRIPTION:
Seventy-two subjects will be randomized into either a traditional landmark-based lumbar puncture or an ultrasound-guided lumbar puncture for obtaining CSF. This study will be conducted in the Neurology clinic. For subjects in the traditional group, the site of needle entry will be determined through palpation of the spine. For subjects in the ultrasound group, site entry will be done using ultrasound guidance. Success and failure of these techniques will be compared along with secondary outcome measures aimed at assessing the safety and efficacy of each of these techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for LP through Neurology's LP clinic
* 18 years of age or older
* Able to understand the description of procedure and provide informed consent

Exclusion Criteria:

* Any contraindications to doing a standard lumbar puncture; which typically includes risk of bleeding from effects of anticoagulants or bleeding disorders or an infection at the potential site of entry in the back. This includes subjects with spinal cord stimulators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Success rate of obtaining CSF within 3 attempts | During the baseline visit, approximately 1 hour
  The success of the procedure is defined as the ability to obtain CSF within 3 attempts via Landmark based LP vs Ultrasound guided LP

SECONDARY OUTCOMES:
Time to completion of LP, in minutes | Immediately following consent, during baseline visit, approximately 1 hour
  Time taken to complete procedure, either traditional vs. ultrasound LP, to obtain CSF
Number of attempts to obtain CSF | Immediately following consent, during baseline visit
  The number of attempts it takes to obtain CSF
Incidence of traumatic tap | Time taken to run analysis of CSF RBC count, approximately within 1 day
  defined as CSF RBC count >400/ml
Pain after the procedure | Immediately post-procedure, approximately 5 minutes
  Universal Pain Assessment Tool: Subject-reported pain level as rated on a scale of 0 - 10. Lower score indicates a better outcome.
Occurrence of post LP headache | Phone call within 72 hours of procedure
  Subject-reported incidence of post LP headache within 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States